CLINICAL TRIAL: NCT02388165
Title: A PHASE 2B, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO EVALUATE THE SAFETY AND EFFICACY OF STAPHYLOCOCCUS AUREUS 4 ANTIGEN VACCINE (SA4AG) IN ADULTS UNDERGOING ELECTIVE OPEN POSTERIOR SPINAL FUSION PROCEDURES WITH MULTILEVEL INSTRUMENTATION
Brief Title: Safety and Efficacy of SA4Ag Vaccine in Adults Having Elective Open Posterior Spinal Fusion Procedures With Multilevel Instrumentation
Acronym: STRIVE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated by sponsor
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B3451002; 2014-002644-40 (EudraCT Number); 6123K1-2001 (Other: Alias Study Number); STRIVE (Other: Alias Study Number)
Record Dates: First submitted 2015-03-09; First posted 2015-03-13 (Estimated); Results first posted 2020-09-02 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-11

CONDITIONS: Staphylococcal Vaccine
Keywords: Staphylococcal Vaccine; Post-operative Surgical Site Infection; Spinal Surgery; MRSA; Staphylococcus aureus
MeSH Terms: conditions — Staphylococcal Infections | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SA4Ag (Active Comparator): Staphylococcus aureus 4-antigen Vaccine
  Interventions: Biological: Staphylococcus aureus 4-Antigen (SA4Ag) Vaccine
- Placebo (Placebo Comparator): Diluent (sterile water) for Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Staphylococcus aureus 4-Antigen (SA4Ag) Vaccine — SA4Ag vaccine reconstituted in 0.5mL water for injection. Administered via IM injection, once 10 to 60 days prior to surgery
  Other Names: Vaccine
  Arms: SA4Ag
Other: Placebo — Vaccine excipients reconstituted in 0.5mL water for injections. Administered via IM injection given 10 to 60 days prior to surgery
  Arms: Placebo

SUMMARY:
The purposes of the clinical trial are to determine whether the SA4Ag vaccine can prevent postoperative Staphylococcus aureus infections in patients who are undergoing elective spinal fusion surgery, and to evaluate the safety of SA4Ag in patients who are undergoing elective spinal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be scheduled to undergo an elective open posterior spinal fusion procedures with multilevel instrumentation, 10 to 60 days after study vaccination.
* Subject must be available for the entire duration of the study, and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures including completion of the electronic diary for 10 days after study vaccination.
* Aged 18 to <86 years old

Exclusion Criteria:

* Planned spinal fusion procedure requiring separate operations performed on separate days (ie, staged procedure).
* Surgical indication of malignancy, infection or acute or emergency trauma.
* History of major surgery within 3 months prior to enrollment, or anticipated major surgery other than the Index Surgical Procedure between study enrollment and completion of study participation.
* History of any spinal surgery performed within 6 months prior to study enrollment.
* History of any previous spinal surgery resulting in postoperative BSI or SSI.
* Congenital or acquired immunodeficiency disorder, rheumatologic disorder or other illness requiring chronic treatment with known immunosuppressant medications, including monoclonal antibodies within a year of enrollment or the use of systemic corticosteroids for > 14 days within 30 days prior to enrollment.
* History of leukemia, lymphoma, underlying bone marrow disorder or history of bone marrow transplant.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3450 (Actual)
Dates: Start 2015-07-02 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (296):
- United States (232):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Brain and Spine, Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Greenbaum Surgical Specialty Hospital, Scottsdale, Arizona
  - HonorHealth Scottsdale Osborn Medical Center, Scottsdale, Arizona
  - Clinical Office - Jason Cuellar M.D., Beverly Hills, California
  - Memorial Orthopaedic Surgical Group, Long Beach, California
  - IDS Pharmacy-USC Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Keck Hospital of USC, Los Angeles, California
  - USC Spine Center, Los Angeles, California
  - USC/Department of Neurological Surgery, Los Angeles, California
  - Cedars-Sinai Medical Center - Investigational Drug, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Clinical Office, Los Angeles, California
  - The Spine Center at Cedars-Sinai, Mark Goodson Building, Cedars-Sinai Medical Center, Los Angeles, California
  - Ronald Reagan Med Center - University of California, Los Angeles (UCLA), Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA CTRC Outpatient Unit, Los Angeles, California
  - Kaiser Permanente Pediatric Clinic, Oakland, California
  - Kaiser Permanente Vaccine Study Center, Oakland, California
  - University of California Irvine Medical Center, Orange, California
  - University of California, San Francisco, San Francisco, California
  - UCLA Spine Center, Santa Monica, California
  - Santa Monica UCLA Medical Center & Orthopaedic Hospital, Santa Monica, California
  - UCLA Santa Monica Infectious Disease, Santa Monica, California
  - LA BioMed at Harbor-UCLA Medical Center, Torrance, California
  - LA BioMed, Harbor-UCLA Medical Center, Torrance, California
  - Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Clinical & Translational Research Center Clinic, Aurora, Colorado
  - University of Colorado Denver, School of Medicine, Aurora, Colorado
  - University of Colorado Department of Pharmacy AIP 2, Pharmacy Bulk Storage, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Health - Foothills Hospital, Boulder, Colorado
  - Boulder Community Health, Boulder, Colorado
  - Justin Parker Neurological Institute, Boulder, Colorado
  - University of Colorado Hospital, Lone Tree Health Center, Lone Tree, Colorado
  - Yale New Haven Hospital - Investigational Drug Services, New Haven, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Yale New Haven Hospital - St. Raphael campus, New Haven, Connecticut
  - Ycci-Csru, New Haven, Connecticut
  - Yale-New Haven Hospital Spine Center, New Haven, Connecticut
  - Holmes Regional Medical Center, Melbourne, Florida
  - The B.A.C.K. Center, Melbourne, Florida
  - Melbourne Regional Medical Center, Melbourne, Florida
  - University of Miami Hospital and Clinics and Research Pharmacy, Miami, Florida
  - University of Miami Hospital, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Neuroscience ACS Research, Orlando, Florida
  - Florida Hospital Orlando - Florida Hospital Investigational Drug Pharmacy, Orlando, Florida
  - Gulfcoast Research Institute, LLC, Sarasota, Florida
  - Emory University Clinic, Atlanta, Georgia
  - Emory Orthopaedics & Spine Center, Atlanta, Georgia
  - Emory Orthopaedics & Spine Hospital, Tucker, Georgia
  - Bingham Memorial Hospital, Blackfoot, Idaho
  - Bingham Memorial Specialty Clinic, Idaho Falls, Idaho
  - Brent H. Greenwald, M.D. Neurological Surgery, Idaho Falls, Idaho
  - Eastern Idaho Regional Medical Center, Idaho Falls, Idaho
  - Mountain View Hospital, Idaho Falls, Idaho
  - Snake River Research, PLLC, Idaho Falls, Idaho
  - Physicians & Surgeons Clinic, Pocatello, Idaho
  - Bingham Memorial Family Medicine & Specialty Clinic, Pocatello, Idaho
  - University of Illinois Hospital and Health Sciences System - Hospital Pharmacy Services, Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System, Chicago, Illinois
  - Rush University Medical Center (RUMC) / Midwest Orthopedics at Rush University Medical Center (RUMC), Chicago, Illinois
  - Rush University Medical Center Pharmacy, Chicago, Illinois
  - Rush University Medical Center Professional Office Building Infusion Pharmacy, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Norton Healthcare Pharmacy, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - Norton Leatherman Spine Center, Louisville, Kentucky
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - AAMC Research Pharmacy, Annapolis, Maryland
  - Anne Arundel Health System Research Institute (AAHSRI), Annapolis, Maryland
  - Anne Arundel Medical Center Infusion Center, Annapolis, Maryland
  - Anne Arundel Medical Center Laboratory, Annapolis, Maryland
  - Anne Arundel Medical Group Orthopedics and Sports Medicine Specialists, Annapolis, Maryland
  - University of Maryland Medical Systems, Department of Neurosurgery, Baltimore, Maryland
  - University of Maryland Medical Systems, Investigational Drug Services, Baltimore, Maryland
  - University of Maryland, Medical Systems, Oriole Park, Baltimore, Maryland
  - John Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Department of Orthopedic Surgery, The Johns Hopkins Outpatient Center, Baltimore, Maryland
  - John Hopkins Hospital, Baltimore, Maryland
  - The Johns Hopkins Hospital Investigational Drug Service, Baltimore, Maryland
  - Anne Arundel Medical Group Orthopedics and Sports Medicine Specialists, Bowie, Maryland
  - Anne Arundel Medical Group Orthopedics and Sports Medicine Specialists, Odenton, Maryland
  - Anne Arundel Medical Group Orthopedics and Sports Medicine Specialists, Pasadena, Maryland
  - Massachusetts General Hospital, Clinical Research Pharmacy, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital Investigational Drug Services (IDS), Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - UMass Memorial Medical Center- Clinical Research Center, Worcester, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Massachusetts Medical Center Memorial Campus, Worcester, Massachusetts
  - University of Michigan Investigational Pharmacy, Ann Arbor, Michigan
  - University Of Michigan Hospitals, Ann Arbor, Michigan
  - Detroit Receiving Hospital, Heart Hospital, Harper Hospital at, Detroit, Michigan
  - Butterworth Hospital, Grand Rapids, Michigan
  - Blodgett Hospital, Grand Rapids, Michigan
  - Orthopaedic Associates of Michigan - Research, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Bronson Spine and Scoliosis Specialists, Kalamazoo, Michigan
  - Michigan Orthopaedic & Spine Surgeons, Rochester Hills, Michigan
  - Beaumont Orthopaedic Center, Royal Oak, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Michigan Orthopaedic Institute, Southfield, Michigan
  - Beaumont Health-Troy, Troy, Michigan
  - Michigan Orthopaedic Institute, West Bloomfield, Michigan
  - Twin Cities Spine Surgeons dba Twin Cities Spine Center, Minneapolis, Minnesota
  - Allina Health - Abbott Northwestern Hospital /, Minneapolis, Minnesota
  - Mayo Clinic Hospital, Methodist Campus, Rochester, Minnesota
  - Mayo Clinic Rochester, Methodist Hospital Campus, Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Center for Outpatient Health, St Louis, Missouri
  - Barnes Jewish Center for Advanced Medicine, St Louis, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - Barnes Jewish Pharmacy, St Louis, Missouri
  - Barnes-Jewish Pharmacy, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - The Rothman Institute Marlton, NJ Office, Marlton, New Jersey
  - HackensackUMC Mountainside Hospital, Montclair, New Jersey
  - Meridian Hospitals Corp c/o Jersey Shore University Medical Center, Neptune City, New Jersey
  - Ambulatory Care Center, Newark, New Jersey
  - Cancer Center, Rutgers, The State University of New Jersey-New Jersey Medical School, Newark, New Jersey
  - Doctors Office Center-Rutgers, The State University of New Jersey-New Jersey Medical School, Newark, New Jersey
  - University Hospital - Pharmacy, Newark, New Jersey
  - University Hospital, Newark, New Jersey
  - The Rothman Institute Washington Township, NJ Office, Sewell, New Jersey
  - Northwell Health Physician Partners- Department of Neurosurgery Spine @Great Neck, Great Neck, New York
  - NYU Langone Huntington Medical Group, Huntington Station, New York
  - UHS Neurosurgery, Johnson City, New York
  - UHS Wilson Medical Center, Johnson City, New York
  - Northwell Health Physician Partners- Department of Neurosurgery Spine @Lynbrook, Lynbrook, New York
  - North Shore University Hospital, Manhasset, New York
  - The Feinstein Institute for Medical Research, Manhasset, New York
  - NYU Langone Health Orthopedic Hospital, New York, New York
  - Kimmel Pavillion, New York, New York
  - NYU Langone Health Orthopedic Center, New York, New York
  - NYU Langone Health Tisch Hospital, New York, New York
  - NYU Langone Madison Ave. Orthopedics, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - lcahn School of Medicine at Mount Sinai, New York, New York
  - The Clinical Research Unit at Mount Sinai, New York, New York
  - NYU Langone Seaport Orthopaedics, New York, New York
  - Carolina Neurosurgery and Spine Associates, P.A., Charlotte, North Carolina
  - Novant Health Charlotte Orthopedic Hospital/Presbyterian Orthopedic Hospital, Charlotte, North Carolina
  - OrthoCarolina Hip & Knee Center, Charlotte, North Carolina
  - OrthoCarolina, Charlotte, North Carolina
  - OrthoCarolina Pineville, Charlotte, North Carolina
  - OrthoCarolina Ballantyne, Charlotte, North Carolina
  - Duke University Hospital, IDS Pharmacy, Durham, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - OrthoCarolina Matthews, Matthews, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - The Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation - Investigation Pharmacy, Cleveland, Ohio
  - Cleveland Clinic Foundation Center for Spine Health, Cleveland, Ohio
  - Riverside Methodist Hospital Pharmacy, Columbus, Ohio
  - Remington-Davis, Inc., Columbus, Ohio
  - Orthopedic One, Columbus, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - OHSU Research Pharmacy, Portland, Oregon
  - Oregon Health and Sciences University, Portland, Oregon
  - Abington Jefferson Health-Pharmacy Department, Abington, Pennsylvania
  - Abington Jefferson Health, Abington, Pennsylvania
  - Rothman Institute-Chalfont Office, Chalfont, Pennsylvania
  - Milton S. Hershey Medical Center Pharmacy, Hershey, Pennsylvania
  - Penn State College of Medicine and Penn State Hershey Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Investigational Drug Service Pharmacy, Philadelphia, Pennsylvania
  - Jefferson Hospital For Neuroscience, Philadelphia, Pennsylvania
  - The Rothman Institute, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital - Pre-Admission Testing Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Cardiovascular Associates, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Upmc (Puh/Muh), Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Rothman Institute-Willow Grove Office, Willow Grove, Pennsylvania
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Austin Infectious Disease Consultants, Austin, Texas
  - Employee Wellness Center, Austin, Texas
  - Seton Medical Center Austin, Austin, Texas
  - St. David's Medical Center, Austin, Texas
  - St. David's Neuroscience and Spine Institute, Austin, Texas
  - Seton Spine and Scoliosis Center, Austin, Texas
  - St. David's North Austin Medical Center, Austin, Texas
  - Wellness Brain and Spine, Austin, Texas
  - Neurosurgical Specialist of Texas, Fredericksburg, Texas
  - Hermann Drive Surgical Hospital, Houston, Texas
  - Mermorial Hermann - Memorial City Medical Center, Houston, Texas
  - Baylor College of Medicine - McNair Campus, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - CHI St. Luke's Health Baylor College of Medicine Medical Center, Houston, Texas
  - Baylor Scott & White Medical Center, Plano, Texas
  - Seton Brain and Spine Institute Williamson, Round Rock, Texas
  - Seton Medical Center Williamson, Round Rock, Texas
  - St. David's Round Rock Medical Center, Round Rock, Texas
  - Scott & White Memorial Hospital and Clinic (Scott & White Roney Bone & Joint Institute), Temple, Texas
  - Scott & White Memorial Hospital and Clinic, Temple, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Clinical Alliance for Research and Education - Infectious Diseases, LLC (CARE-ID), Annandale, Virginia
  - University of Virginia Health System, Charlottesville, Virginia
  - Inova Medical Group, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Inova Neurosciences Research, Falls Church, Virginia
  - OrthoVirginia, McLean, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Sentara Medical Group DBA Sentara Neurosurgery Specialists, Norfolk, Virginia
  - VCU Medical Center Investigational Drug Service, Richamond, Virginia
  - VCU Heatlh Neuroscience Orthopedic and Wellness Center, Richmond, Virginia
  - VCU Health Ambulatory Care Center, Richmond, Virginia
  - VCU Health, Richmond, Virginia
  - Carilion Assessment, Registration and Education for Surgery (C.A.R.E.S), Roanoke, Virginia
  - Carilion Clinic - Department of Pharmacy, Roanoke, Virginia
  - Carilion Clinic Institute for Orthopaedics and Neurosciences, Roanoke, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Carilion Clinic Riverside 3, Roanoke, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - WVU Medicine Spine Center, Morgantown, West Virginia
  - WVU Medicine JW Ruby Memorial Hospital, Morgantown, West Virginia
  - WVU Medicine JW Ruby Memorial Hospital In-Patient Pharmacy, Morgantown, West Virginia
  - WVU Medicine Physician Office Center Orthopaedic Surgery, Morgantown, West Virginia
  - WVU Medicine Physician Office Center, Morgantown, West Virginia
- Austria (2):
  - Tirol Kliniken GmbH, Innsbruck
  - Tirol Kliniken, Innsbruck
- MHAT "Sveta Marina" EAD, Varna, Bulgaria
- Canada (9):
  - Foothills Medical Centre, Calgary, Alberta
  - Foothills Medical Centre, University of Calgary, Calgary, Alberta
  - The Ottawa Hospital, Civic Campus, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - St, Michael's Hospital - St. Michael's Pharmacy, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Montreal Neurological Hospital Research Pharmacy, Montreal, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - Montreal General Hospital Research Institute of the MUHC- MGH Pharmacy Research, Montreal, Quebec
- France (18):
  - CHU Pellegrin Tripode, Bordeaux
  - CHU Pellegrin, Pharmacie, Bordeaux
  - CHU de Dijon, Dijon
  - CHU Hopital d'Enfants, Dijon
  - AP-HM La Timone - Hopital adultes, Marseille
  - AP-HM Hopital Nord, Marseille
  - CHU de Nantes - Hotel Dieu, Nantes
  - CHU de Nimes - Caremeau, Nîmes
  - CHU de Nimes, Nîmes
  - CIC Cochin/Pasteur (CIC 1417), Paris
  - Service de Chirurgie Orthopedique et Traumatologie, Paris
  - Service de Pharmacie, Paris
  - CHU de Rennes - Hopital Pontchaillou, Rennes
  - CHU de Rennes, Rennes
  - Unite d'investigation clinique, Rennes
  - Hopital Nord-CHU Saint Etienne, Saint-Priest-en-Jarez
  - Hopital Civil, Strasbourg
  - Hopitaux Universitaires de Strasbourg, Strasbourg
- Germany (5):
  - Charite- University Medicine Berlin, Berlin
  - Uniklinik Koeln, Cologne
  - Klinikum rechts der Isar, Technische Universitat Munchen, München
  - Klinikum rechts der Isar, München
  - St. Franziskus Hospital Munster, Münster
- Orszagos Gerincgyogyaszati Kozpont, Budapest, Hungary
- Japan (10):
  - Hakodate Central General Hospital, Hakodate, Hokkaido
  - National Hospital Organization Hokkaido Medical Center, Sapporo, Hokkaido
  - Japan Organization of Occupational Health and Safety, Kanto Rosai Hospital, Kawasaki, Kanagawa
  - Nagasaki Rosai Hospital, Sasebo, Nagasaki
  - Saiseikai Kawaguchi General Hospital, Kawaguchi, Saitama
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - National Hospital Organization Murayama Medical Center, Musashimurayama, Tokyo
  - Musashino Red Cross Hospital, Musashino, Tokyo
  - Shimonoseki City Hospital, Shimonoseki-shi, Yamaguchi
  - Japan Community Health care Organization Osaka Hospital, Osaka
- Spain (10):
  - Hospital Clínico Universitario Santiago de Compostela, Santiago de Compostela, A Coruna
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Ramon Y Cajal, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Politecnico La Fe, Valencia
  - Pharmacy Service of Hospital Clinico de Valladolid, Valladolid
  - Hospital Clinico Universitario de Valladolid, Valladolid
- GHP Stockholm Spine Center, Upplands Vasby, Sweden
- United Kingdom (7):
  - Pharmacy Store, Main Pharmacy, Middlesbrough, Cleveland
  - Pharmacy Store, Middlesbrough, Cleveland
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough, Cleveland
  - The James Cook University Hospital, Middlesbrough, Cleveland
  - Salford Royal NHS Foundation Trust, Salford, Greater Manchester
  - Centre for Spinal Studies and Surgery, Nottingham
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Hassanzadeh H, Baber J, Begier E, Noriega DC, Konishi H, Yato Y, Wang MY, Le Huec JC, Patel V, Varga P, Liljenqvist U, Conly J, Sabharwal C, Munjal I, Cooper D, Radley D, Jaques A, Patton M, Gruber WC, Jansen KU, Anderson AS, Gurtman A; STaphylococcus aureus suRgical Inpatient Vaccine Efficacy Investigator Team. Efficacy of a 4-Antigen Staphylococcus aureus Vaccine in Spinal Surgery: The STaphylococcus aureus suRgical Inpatient Vaccine Efficacy (STRIVE) Randomized Clinical Trial. Clin Infect Dis. 2023 Jul 26;77(2):312-320. doi: 10.1093/cid/ciad218. PMID 37125490
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3451002&StudyName=Safety%20and%20Efficacy%20of%20Staphylococcus%20Aureus%204-antigen%2028SA4Ag29%20Vaccine%20in%20Adults%20Undergoing%20Elective%20Posterior%20Instrumented%20Lumbar%20Spinal

RESULTS

PARTICIPANT FLOW:
Groups:
- Staphylococcus Aureus 4-antigen (SA4Ag): Participants randomized to SA4Ag received a single dose of 0.5 milliliter (mL) SA4Ag vaccine intramuscularly, 10 to 60 days prior to their scheduled surgery. Participants were followed from vaccination up to 6 months after their spinal surgical procedure.
- Placebo: Participants randomized to this arm received placebo containing the vaccine excipients reconstituted in 0.5mL water for injection. It was administered via intramuscular injection, 10 to 60 days prior to scheduled surgery. Participants were followed from vaccination up to 6 months after their spinal surgical procedure.
Period: Overall Study
Arm/Group | Staphylococcus Aureus 4-antigen (SA4Ag) | Placebo
Started | 1726 | 1724
Vaccinated (Safety Population) | 1708 | 1709
Completed | 1599 | 1594
Not Completed | 127 | 130
Not completed — Study terminated by sponsor | 5 | 5
Not completed — Other | 11 | 13
Not completed — No longer meet eligibility criteria | 40 | 43
Not completed — Withdrawal of consent | 31 | 32
Not completed — Lost to Follow-up | 19 | 20
Not completed — Death | 13 | 10
Not completed — Adverse Event | 3 | 5
Not completed — Did not meet entrance criteria | 5 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who had received investigational product in this study.
Groups:
- Staphylococcus Aureus 4-antigen (SA4Ag): Participants randomized to SA4Ag received a single dose of 0.5 mL SA4Ag vaccine intramuscularly, 10 to 60 days prior to their scheduled surgery. Participants were followed from vaccination up to 6 months after their spinal surgical procedure.
- Total: Total of all reporting groups
Arm/Group | Staphylococcus Aureus 4-antigen (SA4Ag) | Placebo | Total
Number analyzed (Participants) | 1708 | 1709 | 3417
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (12.3) | 62.6 (12.6) | 62.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 950 | 940 | 1890
  Male | 758 | 769 | 1527
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 69 | 69 | 138
  Not Hispanic or Latino | 1634 | 1639 | 3273
  Unknown or Not Reported | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 295 | 290 | 585
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 90 | 111 | 201
  White | 1295 | 1283 | 2578
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 28 | 25 | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Staphylococcus (S.) Aureus Bloodstream Infection (BSI) And/or Surgical-site Infection (SSI-Including Deep Incisional or Organ/Space) Occurred Within 90 Days After Spinal Surgery
Description: BSI: clinical infection involved a recognized pathogen (S. aureus) cultured from 1 or more blood cultures or a commensal organism cultured from 2 or more blood cultures whether primary or secondary to infection at another site. SSI: infection at a surgical incision. Types of SSI in this outcome measure: Deep incisional SSI: infection involved deep soft tissues of incision (example [e.g.] fascial and muscle layers), Organ/space SSI: infection involved any part of body excluding skin incision, fascia or muscle layers, that was opened or manipulated during operative procedure. Overall number of participants with postoperative BSI and/or SSI (including deep incisional or organ/space), caused by S. aureus, occurred within 90 days of post elective open posterior spinal fusion surgery with multilevel instrumentation, as confirmed by event adjudication committee (EAC) have been reported. A participant may have met criteria for both BSI and SSI (deep incisional or organ/space).
Time Frame: Day of surgery (Day 1) up to Day 90
Population: Per-protocol (PP) efficacy population: all eligible participants, vaccinated as randomized, who underwent surgery per study-defined criteria within 9-90 days (inclusive) post vaccination (expanded from 10-60 days window in protocol), had no infection/malignancy at surgery and had no major protocol violation prior to reporting S. aureus infection.
Measure: Count of Participants; unit: Participants
Arm/Group | Staphylococcus Aureus 4-antigen (SA4Ag) | Placebo
Number analyzed (Participants) | 1544 | 1547
Participants | 14 | 14
Statistical Analysis 1: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Test type: Superiority; Vaccine Efficacy (VE) = 0.00, 95% CI 2-sided [-126.30 to 55.81] — VE was calculated as 1-(P/[1-P]*100), where P is the number of SA4Ag cases divided by the total number of cases. The confidence interval (CI) was calculated using the Clopper-Pearson method

2. Primary Outcome: Percentage of Participants With Local Reactions Within 10 Days After Vaccination
Description: Local reactions were recorded using an electronic diary (e-diary). Local reactions included redness, swelling and pain at the injection site. Redness and swelling were categorized as mild (2.5 to 5.0 centimeters [cm]), moderate (5.5 to 10.0 cm) and, severe (greater than or equal to [>=] 10.5 cm). Pain at the injection site was defined as mild (did not interfere with activity), moderate (interfered with activity), and severe (prevented daily activity). Participants may be represented in more than 1 row. Here, "Any" for redness, swelling, pain at the injection site represents any grade of these local reactions among mild, moderate or severe.
Time Frame: Within 10 days after Vaccination
Population: Safety population: all participants who received investigational product in this study. Here, "Overall Number of Participants Analyzed, N" signifies number of participants analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Staphylococcus Aureus 4-antigen (SA4Ag) | Placebo
Number analyzed (Participants) | 1692 | 1685
Percentage of participants
  Redness: Any | 9.2 [7.9 to 10.7] | 0.9 [0.5 to 1.5]
  Redness: Mild | 5.3 [4.2 to 6.4] | 0.9 [0.5 to 1.5]
  Redness: Moderate | 3.1 [2.4 to 4.1] | 0.1 [0.0 to 0.3]
  Redness: Severe | 0.8 [0.5 to 1.4] | 0.0 [0.0 to 0.2]
  Swelling: Any | 8.0 [6.7 to 9.4] | 1.0 [0.6 to 1.6]
  Swelling: Mild | 4.6 [3.6 to 5.7] | 0.7 [0.4 to 1.2]
  Swelling: Moderate | 2.7 [2.0 to 3.6] | 0.3 [0.1 to 0.7]
  Swelling: Severe | 0.7 [0.4 to 1.2] | 0.0 [0.0 to 0.2]
  Pain at the injection site: Any | 24.1 [22.1 to 26.2] | 8.4 [7.1 to 9.9]
  Pain at the injection site: Mild | 19.2 [17.4 to 21.2] | 7.0 [5.8 to 8.3]
  Pain at the injection site: Moderate | 4.3 [3.4 to 5.4] | 1.3 [0.8 to 2.0]
  Pain at the injection site: Severe | 0.6 [0.3 to 1.1] | 0.1 [0.0 to 0.4]
Statistical Analysis 1: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Redness: Any; Test type: Superiority; p < 0.001, Miettinen and Nurminen; Difference in percentage of participants = 8.3, 95% CI 2-sided [6.9 to 9.8]
Statistical Analysis 2: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Redness: Mild; Test type: Superiority; Difference in percentage of participants = 4.4, 95% CI 2-sided [3.3 to 5.6]
Statistical Analysis 3: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Redness: Moderate; Test type: Superiority; Difference in percentage of participants = 3.0, 95% CI 2-sided [2.3 to 4.0]
Statistical Analysis 4: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Redness: Severe; Test type: Superiority; Difference in percentage of participants = 0.8, 95% CI 2-sided [0.5 to 1.4]
Statistical Analysis 5: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Swelling: Any; Test type: Superiority; p < 0.001, Miettinen and Nurminen; Difference in percentage of participants = 7.0, 95% CI 2-sided [5.7 to 8.4]
Statistical Analysis 6: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Swelling: Mild; Test type: Superiority; Difference in percentage of participants = 3.9, 95% CI 2-sided [2.8 to 5.0]
Statistical Analysis 7: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Swelling: Moderate; Test type: Superiority; Difference in percentage of participants = 2.4, 95% CI 2-sided [1.7 to 3.3]
Statistical Analysis 8: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Swelling: Severe; Test type: Superiority; Difference in percentage of participants = 0.7, 95% CI 2-sided [0.4 to 1.2]
Statistical Analysis 9: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Pain at the injection site: Any; Test type: Superiority; p < 0.001, Miettinen and Nurminen; Difference in percentage of participants = 15.7, 95% CI 2-sided [13.3 to 18.1]
Statistical Analysis 10: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Pain at the injection site: Mild; Test type: Superiority; Difference in percentage of participants = 12.2, 95% CI 2-sided [10.0 to 14.5]
Statistical Analysis 11: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Pain at the injection site: Moderate; Test type: Superiority; Difference in percentage of participants = 3.0, 95% CI 2-sided [1.9 to 4.2]
Statistical Analysis 12: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Pain at the injection site: Severe; Test type: Superiority; Difference in percentage of participants = 0.5, 95% CI 2-sided [0.1 to 1.0]

3. Primary Outcome: Percentage of Participants With Systemic Reactions Within 10 Days After Vaccination
Description: Systemic reactions included fever, fatigue, headache, diarrhea, vomiting, muscle pain and joint pain, were recorded using an e-diary. Fever was graded as 38.0 to 38.4 degree Celsius (C), 38.5 to 38.9 degree C, 39.0 to 40.0 degree C and greater than (>) 40.0 degree C. Vomiting was graded as mild (1-2 times in 24 hours), moderate (>2 times in 24 hours) and severe (required intravenous hydration). Diarrhea was graded as mild (2-3 loose stools in 24 hours), moderate (4-5 loose stools in 24 hours) and severe (>=6 loose stools in 24 hours). Headache, fatigue, muscle pain and joint pain were graded as mild (no interference with activity), moderate (some interference with activity) and severe (prevented daily routine activity). Participants may be represented in more than 1 row. Here "any" for fever, fatigue, headache, vomiting, diarrhea, muscle pain, joint pain represents any grade of these systemic reactions among mild, moderate or severe.
Time Frame: Within 10 days after Vaccination
Population: Safety population: all participants who received investigational product in this study. Here, "Overall Number of Participants Analyzed" signifies number of participants analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Staphylococcus Aureus 4-antigen (SA4Ag) | Placebo
Number analyzed (Participants) | 1692 | 1685
Percentage of participants
  Fever: Any | 2.0 [1.4 to 2.8] | 1.4 [0.9 to 2.0]
  Fever: 38.0 degree C to 38.4 degree C | 1.3 [0.8 to 2.0] | 0.9 [0.5 to 1.5]
  Fever: 38.5 degree C to 38.9 degree C | 0.5 [0.2 to 0.9] | 0.4 [0.2 to 0.9]
  Fever: 39.0 degree C to 40.0 degree C | 0.2 [0.0 to 0.5] | 0.1 [0.0 to 0.3]
  Fever: >40.0 degree C | 0.1 [0.0 to 0.3] | 0.0 [0.0 to 0.2]
  Fatigue: Any | 43.3 [40.9 to 45.7] | 40.4 [38.1 to 42.8]
  Fatigue: Mild | 14.0 [12.4 to 15.8] | 12.6 [11.1 to 14.3]
  Fatigue: Moderate | 24.9 [22.8 to 27.0] | 23.6 [21.6 to 25.7]
  Fatigue: Severe | 4.4 [3.4 to 5.5] | 4.2 [3.3 to 5.2]
  Headache: Any | 32.4 [30.2 to 34.7] | 31.2 [29.0 to 33.5]
  Headache: Mild | 17.7 [15.9 to 19.6] | 18.0 [16.2 to 19.9]
  Headache: Moderate | 13.5 [11.9 to 15.3] | 12.0 [10.5 to 13.6]
  Headache: Severe | 1.2 [0.8 to 1.9] | 1.2 [0.8 to 1.9]
  Diarrhea: Any | 17.0 [15.2 to 18.8] | 16.0 [14.3 to 17.9]
  Diarrhea: Mild | 13.0 [11.4 to 14.7] | 12.2 [10.7 to 13.9]
  Diarrhea: Moderate | 3.4 [2.6 to 4.4] | 2.9 [2.2 to 3.8]
  Diarrhea: Severe | 0.5 [0.2 to 1.0] | 0.9 [0.5 to 1.5]
  Vomiting: Any | 2.7 [1.9 to 3.5] | 3.3 [2.5 to 4.2]
  Vomiting: Mild | 2.4 [1.7 to 3.2] | 2.6 [1.9 to 3.5]
  Vomiting: Moderate | 0.3 [0.1 to 0.7] | 0.7 [0.3 to 1.2]
  Vomiting: Severe | 0.0 [0.0 to 0.2] | 0.0 [0.0 to 0.2]
  Muscle pain: Any | 27.9 [25.8 to 30.1] | 26.2 [24.1 to 28.4]
  Muscle pain: Mild | 10.1 [8.7 to 11.6] | 9.3 [8.0 to 10.8]
  Muscle pain: Moderate | 15.7 [14.0 to 17.5] | 14.6 [12.9 to 16.4]
  Muscle pain: Severe | 2.1 [1.5 to 2.9] | 2.3 [1.7 to 3.2]
  Joint pain: Any | 27.5 [25.4 to 29.7] | 25.8 [23.7 to 28.0]
  Joint pain: Mild | 9.6 [8.3 to 11.1] | 8.0 [6.7 to 9.3]
  Joint pain: Moderate | 16.1 [14.4 to 17.9] | 16.1 [14.4 to 18.0]
  Joint pain: Severe | 1.8 [1.2 to 2.5] | 1.7 [1.2 to 2.5]
Statistical Analysis 1: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Fever: Any; Test type: Superiority; p = 0.146, Miettinen and Nurminen; Difference in percentage of participants = 0.6, 95% CI 2-sided [-0.2 to 1.6]
Statistical Analysis 2: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Fever: 38.0 degree C to 38.4 degree C; Test type: Superiority; Difference in percentage of participants = 0.4, 95% CI 2-sided [-0.3 to 1.2]
Statistical Analysis 3: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Fever: 38.5 degree C to 38.9 degree C; Test type: Superiority; Difference in percentage of participants = 0.1, 95% CI 2-sided [-0.4 to 0.6]
Statistical Analysis 4: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Fever: 39.0 degree C to 40.0 degree C; Test type: Superiority; Difference in percentage of participants = 0.1, 95% CI 2-sided [-0.2 to 0.5]
Statistical Analysis 5: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Fever: >40.0 degree C; Test type: Superiority; Difference in percentage of participants = 0.1, 95% CI 2-sided [-0.2 to 0.3]
Statistical Analysis 6: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Fatigue: Any; Test type: Superiority; p = 0.093, Miettinen and Nurminen; Difference in percentage of participants = 2.9, 95% CI [-0.5 to 6.2]
Statistical Analysis 7: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Fatigue: Mild; Test type: Superiority; Difference in percentage of participants = 1.4, 95% CI 2-sided [-0.9 to 3.7]
Statistical Analysis 8: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Fatigue: Moderate; Test type: Superiority; Difference in percentage of participants = 1.3, 95% CI 2-sided [-1.6 to 4.2]
Statistical Analysis 9: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Fatigue: Severe; Test type: Superiority; Difference in percentage of participants = 0.2, 95% CI 2-sided [-1.2 to 1.6]
Statistical Analysis 10: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Headache: Any; Test type: Superiority; p = 0.443, Miettinen and Nurminen; Difference in percentage of participants = 1.2, 95% CI 2-sided [-1.9 to 4.4]
Statistical Analysis 11: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Headache: Mild; Test type: Superiority; Difference in percentage of participants = -0.3, 95% CI 2-sided [-2.9 to 2.3]
Statistical Analysis 12: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Headache: Moderate; Test type: Superiority; Difference in percentage of participants = 1.5, 95% CI 2-sided [-0.7 to 3.8]
Statistical Analysis 13: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Headache: Severe; Test type: Superiority; Difference in percentage of participants = 0.0, 95% CI 2-sided [-0.8 to 0.8]
Statistical Analysis 14: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Diarrhea: Any; Test type: Superiority; p = 0.462, Miettinen and Nurminen; Difference in percentage of participants = 1.0, 95% CI 2-sided [-1.6 to 3.4]
Statistical Analysis 15: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Diarrhea: Mild; Test type: Superiority; Difference in percentage of participants = 0.8, 95% CI 2-sided [-1.5 to 3.0]
Statistical Analysis 16: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Diarrhea: Moderate; Test type: Superiority; Difference in percentage of participants = 0.5, 95% CI [-0.7 to 1.7]
Statistical Analysis 17: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Diarrhea: Severe; Test type: Superiority; Difference in percentage of participants = -0.4, 95% CI 2-sided [-1.0 to 0.2]
Statistical Analysis 18: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Vomiting: Any; Test type: Superiority; p = 0.300, Miettinen and Nurminen; Difference in percentage of participants = -0.6, 95% CI [-1.8 to 0.5]
Statistical Analysis 19: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Vomiting: Mild; Test type: Superiority; Difference in percentage of participants = -0.2, 95% CI 2-sided [-1.3 to 0.8]
Statistical Analysis 20: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Vomiting: Moderate; Test type: Superiority; Difference in percentage of participants = -0.4, 95% CI [-0.9 to 0.1]
Statistical Analysis 21: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Muscle pain: Any; Test type: Superiority; p = 0.276, Miettinen and Nurminen; Difference in percentage of participants = 1.7, 95% CI [-1.3 to 4.7]
Statistical Analysis 22: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Muscle pain: Mild; Test type: Superiority; Difference in percentage of participants = 0.8, 95% CI 2-sided [-1.2 to 2.8]
Statistical Analysis 23: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Muscle pain: Moderate; Test type: Superiority; Difference in percentage of participants = 1.1, 95% CI 2-sided [-1.4 to 3.5]
Statistical Analysis 24: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Muscle pain: Severe; Test type: Superiority; Difference in percentage of participants = -0.2, 95% CI [-1.2 to 0.8]
Statistical Analysis 25: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Joint pain: Any; Test type: Superiority; p = 0.273, Miettinen and Nurminen; Difference in percentage of participants = 1.7, 95% CI 2-sided [-1.3 to 4.6]
Statistical Analysis 26: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Joint pain: Mild; Test type: Superiority; Difference in percentage of participants = 1.6, 95% CI 2-sided [-0.2 to 3.6]
Statistical Analysis 27: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Joint pain: Moderate; Test type: Superiority; Difference in percentage of participants = 0.0, 95% CI 2-sided [-2.6 to 2.4]
Statistical Analysis 28: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Joint pain: Severe; Test type: Superiority; Difference in percentage of participants = 0.1, 95% CI [-0.9 to 1.0]

4. Primary Outcome: Number of Participants With Adverse Events (AEs) From Vaccination Until The Day of Surgery (Day 1)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study vaccine without regard to possibility of causal relationship. AEs including serious as well non-serious AEs.
Time Frame: From vaccination up to Day of surgery (Day 1) (10-60 days after vaccination)
Population: Safety population: all participants who received investigational product in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Staphylococcus Aureus 4-antigen (SA4Ag) | Placebo
Number analyzed (Participants) | 1708 | 1709
Participants | 213 | 178

5. Primary Outcome: Number of Participants With Adverse Events (AEs) From Vaccination Until First Postoperative Evaluation on Day 42
Description: An AE was any untoward medical occurrence in a participant who received study vaccine without regard to possibility of causal relationship. AEs including serious as well non-serious AEs.
Time Frame: From vaccination until Day 42 after surgery (52-102 days after vaccination)
Population: Safety population: all participants who received investigational product in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Staphylococcus Aureus 4-antigen (SA4Ag) | Placebo
Number analyzed (Participants) | 1708 | 1709
Participants | 1198 | 1213

6. Primary Outcome: Number of Participants With Adverse Events (AEs) From The Day of Surgery (Day 1) Until First Postoperative Evaluation on Day 42
Description: as for outcome 5
Time Frame: Day of surgery (Day 1) up to Day 42 after surgery
Population: Safety population: all participants who received investigational product in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Staphylococcus Aureus 4-antigen (SA4Ag) | Placebo
Number analyzed (Participants) | 1708 | 1709
Participants | 1136 | 1167

7. Primary Outcome: Number of Participants With Newly Diagnosed Chronic Medical Disorders From First Postoperative Evaluation on Day 42 Until Last Postoperative Evaluation on Day 180
Description: A newly diagnosed chronic medical disorder was defined as a disease or medical condition, not previously identified, that was expected to be persistent or otherwise long-lasting in its effects.
Time Frame: Day 42 up to Day 180 (up to 138 days)
Population: Safety population: all participants who received investigational product in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Staphylococcus Aureus 4-antigen (SA4Ag) | Placebo
Number analyzed (Participants) | 1708 | 1709
Participants | 29 | 41

8. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) From Vaccination Until Last Postoperative Evaluation on Day 180
Description: An AE was any untoward medical occurrence in a participant who received study vaccine without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability/incapacity, congenital anomaly.
Time Frame: From vaccination up to Day 180 after surgery (190-240 days after vaccination)
Population: Safety population: all participants who received investigational product in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Staphylococcus Aureus 4-antigen (SA4Ag) | Placebo
Number analyzed (Participants) | 1708 | 1709
Participants | 403 | 424

9. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) From Vaccination Until Day of Surgery (Day 1)
Description: An AE was any untoward medical occurrence in a participant who received study vaccine without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability/incapacity, congenital anomaly.
Time Frame: From vaccination up to Day of surgery (Day 1) (10-60 days after vaccination)
Population: Safety population: all participants who received investigational product in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Staphylococcus Aureus 4-antigen (SA4Ag) | Placebo
Number analyzed (Participants) | 1708 | 1709
Participants | 27 | 26

10. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) From The Day of Surgery (Day 1) Until Last Postoperative Evaluation on Day 180
Description: as for outcome 9
Time Frame: Day of surgery (Day 1) up to Day 180 after surgery
Population: Safety population: all participants who received investigational product in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Staphylococcus Aureus 4-antigen (SA4Ag) | Placebo
Number analyzed (Participants) | 1708 | 1709
Participants | 384 | 401

11. Secondary Outcome: Number of Participants With Postoperative S. Aureus Blood Stream Infection (BSI) And/or Surgical-site Infection (SSI-Including Deep Incisional or Organ/Space) Occurred Within 180 Days After Surgery
Description: BSI: clinical infection involved a recognized pathogen (S. aureus) cultured from 1 or more blood cultures or a commensal organism cultured from 2 or more blood cultures whether primary or secondary to infection at another site. SSI: infection at a surgical incision. Types of SSI in this outcome measure: Deep incisional SSI: infection involved deep soft tissues of incision (e.g. fascial and muscle layers), Organ/space SSI: infection involved any part of body excluding skin incision, fascia or muscle layers, that was opened or manipulated during operative procedure. Overall number of participants with postoperative BSI and/or SSI (including deep incisional or organ/space), caused by S. aureus, occurred within 180 days of post elective open posterior spinal fusion surgery with multilevel instrumentation, as confirmed by EAC have been reported. A participant may have met criteria for both BSI and SSI (deep incisional or organ/space).
Time Frame: Day of surgery (Day 1) up to Day 180 after surgery
Population: PP efficacy population: all eligible participants, vaccinated as randomized, who underwent surgery per study-defined criteria within 9-90 days (inclusive) post vaccination (expanded from 10-60 days window in protocol), had no infection/malignancy at surgery and had no major protocol violation prior to reporting S. aureus infection.
Measure: Count of Participants; unit: Participants
Arm/Group | Staphylococcus Aureus 4-antigen (SA4Ag) | Placebo
Number analyzed (Participants) | 1544 | 1547
Participants | 14 | 14
Statistical Analysis 1: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Test type: Superiority; VE = 0.0, 95% CI 2-sided [-126.30 to 55.81] — VE was calculated as 1-(P/[1-P]*100), where P is the number of SA4Ag cases divided by the total number of cases. The CI was calculated using the Clopper-Pearson method

12. Secondary Outcome: Number of Participants With Any Postoperative S. Aureus Surgical-site Infection (SSI-Superficial, Deep Incisional or Organ/Space) Occurred Within 90 Days After Surgery
Description: SSI: infection at a surgical incision. Types of SSI in this outcome measure: Superficial SSI: Infection involved only skin and subcutaneous tissue of the incision, Deep incisional SSI: infection involved deep soft tissues of incision (e.g. fascial and muscle layers), Organ/space SSI: infection involved any part of body, excluding skin incision, fascia, or muscle layers, that was opened or manipulated during operative procedure. Overall number of participants with postoperative SSI (including superficial, deep incisional and/or organ/space SSI) caused by S. aureus, occurred within 90 days after elective open posterior spinal fusion surgery with multilevel instrumentation as confirmed by EAC have been reported.
Time Frame: Day of surgery (Day 1) up to Day 90 after surgery
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Staphylococcus Aureus 4-antigen (SA4Ag) | Placebo
Number analyzed (Participants) | 1544 | 1547
Participants | 24 | 22
Statistical Analysis 1: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Test type: Superiority; VE = -9.09, 95% CI 2-sided [-104.06 to 41.41] — [estimate comment as in outcome 11, analysis 1]

13. Secondary Outcome: Number of Participants With Any Postoperative S. Aureus Surgical-site Infection (SSI-Superficial, Deep Incisional or Organ/Space) Occurred Within 180 Days After Surgery
Description: SSI: infection at a surgical incision. Types of SSI in this outcome measure: Superficial SSI: Infection involved only skin and subcutaneous tissue of the incision, Deep incisional SSI: infection involved deep soft tissues of incision (e.g. fascial and muscle layers), Organ/space SSI: infection involved any part of body, excluding skin incision, fascia, or muscle layers, that was opened or manipulated during operative procedure. Overall number of participants with postoperative SSI (including superficial, deep incisional and/or organ/space SSI) caused by S. aureus, occurred within 180 days after elective open posterior spinal fusion surgery with multilevel instrumentation as confirmed by EAC have been reported.
Time Frame: Day of surgery (Day 1) up to Day 180 after surgery
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Staphylococcus Aureus 4-antigen (SA4Ag) | Placebo
Number analyzed (Participants) | 1544 | 1547
Participants | 25 | 23
Statistical Analysis 1: Comparison: Staphylococcus Aureus 4-antigen (SA4Ag) vs Placebo; Test type: Superiority; VE = -8.70, 95% CI 2-sided [-100.42 to 40.80] — [estimate comment as in outcome 11, analysis 1]

ADVERSE EVENTS:
Time Frame: SAE and non-SAE: From vaccination up to Day 180 (190-240 days after vaccination). Local and systemic reactions: within 10 days after vaccination (systematic assessment).
Description: Safety population: included all participants who had received investigational product in this study. The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant or one participant may have experienced both a serious and non-serious event during the analysis population.
Arm/Group | Staphylococcus Aureus 4-antigen (SA4Ag) | Placebo
All-Cause Mortality (participants affected / at risk) | 13/1708 | 10/1709
Serious Adverse Events (participants affected / at risk) | 403/1708 | 424/1709
Other Adverse Events (participants affected / at risk) | 1530/1708 | 1489/1709
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Staphylococcus Aureus 4-antigen (SA4Ag) (N=1708) | Placebo (N=1709)
Anaemia (Blood and lymphatic system disorders) | 4 | 4
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Platelet disorder (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 3 | 4
Acute right ventricular failure (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 1 | 0
Arteriospasm coronary (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 12 | 10
Atrial flutter (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 2 | 2
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 4
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 2 | 0
Coronary artery disease (Cardiac disorders) | 1 | 4
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 2
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 4 | 2
Sinus node dysfunction (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 2 | 3
Ventricular tachycardia (Cardiac disorders) | 0 | 2
Spinal muscular atrophy (Congenital, familial and genetic disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 2
Retinal detachment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 1
Anorectal disorder (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 2
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 2 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 2 | 5
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 3 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Obstruction gastric (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 3
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Rectal prolapse (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Calcinosis (General disorders) | 1 | 0
Chest pain (General disorders) | 3 | 5
Complication associated with device (General disorders) | 0 | 2
Complication of device insertion (General disorders) | 0 | 1
Dysplasia (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
Fibrosis (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
Hernia (General disorders) | 0 | 1
Impaired healing (General disorders) | 2 | 1
Medical device site reaction (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 4 | 3
Pain (General disorders) | 3 | 3
Peripheral swelling (General disorders) | 2 | 1
Pyrexia (General disorders) | 6 | 7
Surgical failure (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 4 | 4
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 2 | 2
Abscess jaw (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 3
Bacterial disease carrier (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 2
Cellulitis (Infections and infestations) | 5 | 4
Clostridium colitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 2
Diverticulitis (Infections and infestations) | 2 | 1
Encephalitis (Infections and infestations) | 1 | 0
Enterobacter bacteraemia (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Extradural abscess (Infections and infestations) | 0 | 1
Fournier's gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Incision site abscess (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 1
Intervertebral discitis (Infections and infestations) | 1 | 2
Lice infestation (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 0
Medical device site joint infection (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 2 | 2
Osteomyelitis chronic (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 19 | 12
Pneumonia bacterial (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 1
Postoperative wound infection (Infections and infestations) | 27 | 32
Pyelonephritis (Infections and infestations) | 2 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 11 | 10
Septic shock (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 0 | 3
Staphylococcal infection (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 6 | 7
Urosepsis (Infections and infestations) | 2 | 1
Viral infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 5 | 5
Wound infection bacterial (Infections and infestations) | 1 | 3
Wound infection fungal (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 3
Adjacent segment degeneration (Injury, poisoning and procedural complications) | 1 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 8 | 3
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2
Aortic injury (Injury, poisoning and procedural complications) | 1 | 0
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1
Concussion (Injury, poisoning and procedural complications) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Device deployment issue (Injury, poisoning and procedural complications) | 1 | 1
Device dispensing error (Injury, poisoning and procedural complications) | 0 | 1
Dural tear (Injury, poisoning and procedural complications) | 9 | 9
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 | 1
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 4 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 9 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 2
Flatback syndrome (Injury, poisoning and procedural complications) | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 3
Graft complication (Injury, poisoning and procedural complications) | 0 | 1
Heart injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Incision site haematoma (Injury, poisoning and procedural complications) | 0 | 1
Incomplete spinal fusion (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 6 | 5
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 3
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural constipation (Injury, poisoning and procedural complications) | 1 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 3 | 2
Post procedural fever (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 3 | 7
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Postoperative delirium (Injury, poisoning and procedural complications) | 1 | 3
Postoperative ileus (Injury, poisoning and procedural complications) | 3 | 7
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 4 | 3
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 7 | 9
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
Seroma (Injury, poisoning and procedural complications) | 6 | 4
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 6 | 2
Spinal cord injury cauda equina (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Suture rupture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 4 | 4
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1
Urethral injury (Injury, poisoning and procedural complications) | 1 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 1
Vascular injury (Injury, poisoning and procedural complications) | 1 | 0
Venous injury (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 5 | 4
Wound secretion (Injury, poisoning and procedural complications) | 1 | 2
Blood glucose increased (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 2
Oxygen saturation decreased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 2
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 3 | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 7
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 3
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 3
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal deformity (Musculoskeletal and connective tissue disorders) | 2 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal instability (Musculoskeletal and connective tissue disorders) | 5 | 3
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal segmental dysfunction (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 3 | 2
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant neoplasm of ampulla of vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 1
Cerebrospinal fistula (Nervous system disorders) | 0 | 2
Cerebrospinal fluid leakage (Nervous system disorders) | 5 | 5
Cerebrovascular accident (Nervous system disorders) | 2 | 2
Cervical radiculopathy (Nervous system disorders) | 2 | 0
Cervical spinal cord paralysis (Nervous system disorders) | 1 | 2
Decreased vibratory sense (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 4 | 5
Facial paralysis (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 2
Hemiparesis (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
IIIrd nerve paresis (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 2
Metabolic encephalopathy (Nervous system disorders) | 1 | 2
Miller Fisher syndrome (Nervous system disorders) | 1 | 0
Monoparesis (Nervous system disorders) | 1 | 1
Monoplegia (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Normal pressure hydrocephalus (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 2
Paralysis (Nervous system disorders) | 3 | 0
Paraparesis (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 2 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 2 | 1
Radiculopathy (Nervous system disorders) | 2 | 2
Sciatica (Nervous system disorders) | 2 | 4
Sedation (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 3 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Spinal cord disorder (Nervous system disorders) | 0 | 1
Spinal epidural haematoma (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 2 | 5
Thalamus haemorrhage (Nervous system disorders) | 1 | 0
Thrombotic cerebral infarction (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 4 | 4
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Visual field defect (Nervous system disorders) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Device breakage (Product Issues) | 2 | 2
Device dislocation (Product Issues) | 11 | 6
Device failure (Product Issues) | 3 | 6
Device fastener issue (Product Issues) | 3 | 1
Device loosening (Product Issues) | 3 | 2
Implant subsidence (Product Issues) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 2
Delirium (Psychiatric disorders) | 3 | 4
Delirium tremens (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 4 | 7
Suicidal ideation (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 6 | 8
Bladder disorder (Renal and urinary disorders) | 1 | 0
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 1
Nephropathy (Renal and urinary disorders) | 0 | 1
Neurogenic bladder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 2
Renal injury (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 4 | 3
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Prostatic haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 22 | 17
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 2
Arthrodesis (Surgical and medical procedures) | 1 | 0
Muscle flap operation (Surgical and medical procedures) | 1 | 0
Spinal fusion surgery (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 21 | 19
Haematoma (Vascular disorders) | 2 | 3
Haemodynamic instability (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 13 | 10
Hypovolaemic shock (Vascular disorders) | 1 | 3
Iliac artery occlusion (Vascular disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 1
Ischaemia (Vascular disorders) | 0 | 1
Labile blood pressure (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 1
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 3 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 2 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Uncoded System Organ Class (Infections and infestations) | 0 | 1
Meningoencephalitis septic shock (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Staphylococcus Aureus 4-antigen (SA4Ag) (N=1708) | Placebo (N=1709)
Anaemia (Blood and lymphatic system disorders) | 97 | 122
Blood loss anaemia (Blood and lymphatic system disorders) | 58 | 42
Leukocytosis (Blood and lymphatic system disorders) | 18 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 26 | 23
Tachycardia (Cardiac disorders) | 32 | 30
Constipation (Gastrointestinal disorders) | 201 | 192
Diarrhoea 1 (Gastrointestinal disorders) | 31 | 30
Nausea (Gastrointestinal disorders) | 162 | 140
Vomiting 1 (Gastrointestinal disorders) | 80 | 67
Chest pain (General disorders) | 18 | 13
Oedema peripheral (General disorders) | 22 | 29
Pyrexia 1 (General disorders) | 121 | 114
Nasopharyngitis (Infections and infestations) | 28 | 23
Urinary tract infection (Infections and infestations) | 96 | 103
Anaemia postoperative (Injury, poisoning and procedural complications) | 109 | 108
Dural tear (Injury, poisoning and procedural complications) | 60 | 73
Fall (Injury, poisoning and procedural complications) | 60 | 44
Incision site pain (Injury, poisoning and procedural complications) | 67 | 63
Procedural pain (Injury, poisoning and procedural complications) | 92 | 84
Wound complication (Injury, poisoning and procedural complications) | 19 | 21
Hyperglycaemia (Metabolism and nutrition disorders) | 28 | 25
Hypokalaemia (Metabolism and nutrition disorders) | 24 | 18
Hyponatraemia (Metabolism and nutrition disorders) | 22 | 20
Arthralgia 1 (Musculoskeletal and connective tissue disorders) | 27 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 39 | 36
Muscle spasms (Musculoskeletal and connective tissue disorders) | 21 | 30
Muscular weakness (Musculoskeletal and connective tissue disorders) | 25 | 24
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 24 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 55 | 59
Dizziness (Nervous system disorders) | 30 | 35
Headache 1 (Nervous system disorders) | 33 | 26
Hypoaesthesia (Nervous system disorders) | 50 | 38
Paraesthesia (Nervous system disorders) | 24 | 12
Insomnia (Psychiatric disorders) | 68 | 63
Acute kidney injury (Renal and urinary disorders) | 24 | 13
Urinary retention (Renal and urinary disorders) | 58 | 59
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 10 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 19
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 24 | 35
Erythema (Skin and subcutaneous tissue disorders) | 57 | 61
Pruritus (Skin and subcutaneous tissue disorders) | 27 | 33
Rash (Skin and subcutaneous tissue disorders) | 21 | 15
Hypertension (Vascular disorders) | 15 | 20
Hypotension (Vascular disorders) | 79 | 84
Diarrhoea 2 (Gastrointestinal disorders) | 287 | 270
Vomiting 2 (Gastrointestinal disorders) | 45 | 55
Fatigue (General disorders) | 732 | 681
Injection site erythema (General disorders) | 156 | 16
Injection site pain (General disorders) | 408 | 142
Injection site swelling (General disorders) | 135 | 17
Pyrexia 2 (General disorders) | 34 | 23
Arthralgia 2 (Musculoskeletal and connective tissue disorders) | 465 | 435
Myalgia (muscle pain) (Musculoskeletal and connective tissue disorders) | 472 | 442
Headache 2 (Nervous system disorders) | 549 | 526

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT02388165/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT02388165/SAP_001.pdf